CLINICAL TRIAL: NCT01507129
Title: Biomarkers for Noninvasive Assessment of Human Hydration
Status: Completed | Type: Observational
Sponsor: Gaia Medical Institute (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: DM102745
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Dehydration
Keywords: dehydration; plasma; osmolality; saliva; urine; biomarkers; hypertonic; isotonic; hydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Serum, Urine, Saliva
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Low levels of dehydration (the loss of body water corresponding to 2% of the body weight), deteriorate physical and cognitive performance and may also be linked to a number of chronic diseases. The standard test used for the assessment of hydration status is plasma osmolality. This blood test is invasive, requires time and laboratory equipment and is not accurate for isotonic dehydration. The goal of this project is to determine whether a new molecular technology, saliva-based Stress Response Profiling (SRP) biomarkers, could be used for non-invasive diagnostics of dehydration.

DETAILED DESCRIPTION:
Dehydration, or the loss of body water, is a common health problem during military operations, athletic events and illness, particularly in children and the elderly. Warfighters frequently become dehydrated when training or fighting in hot and mountainous environments because heat and high altitude increase body water losses. The negative consequences of dehydration worsen as body water losses increase. Severe dehydration (>10%) is a life-threatening emergency that may result in heat illness, seizures, permanent brain damage or death. The most common type of dehydration is caused by sweat loss during heavy physical labor or exercise (hypertonic dehydration). A different type of dehydration can be caused by blood loss, burns, diarrhea, vomiting or diuretic drugs used for example by diabetics (isotonic dehydration). Despite the critical importance of proper fluid balance to human performance and health, no field-expedient, non-invasive dehydration test is available for either form of dehydration. The ultimate goal of this project is to develop a field-expedient, non-invasive test for both types of dehydration. The test will be sensitive to 2% dehydration, a critical threshold for performance impairment and a statistically valid decision point for hydration assessment.

Design: Fifteen volunteers will be first euhydrated (well-hydrated) and then moderately dehydrated (2-4%) using two procedures. First, sweat loss during exercise in the heat without fluids (hypertonic dehydration). Second, excessive urination stimulated by a diuretic pill called Lasix (isotonic dehydration). SRP biomarkers in saliva samples will be compared to changes in body weight, and to known hydration indicators in blood and urine. Results will identify the best SRP biomarkers for diagnosing both types of dehydration and compare accuracy of the new saliva test to the existing hydration indicators.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Males and females between 18-40, healthy and aerobically fit determined by VO2max test. Minimum 45 ml/kg/min for males and 40 ml/kg/min for females
* Willing to stop drinking any alcoholic beverages, taking all supplements and limit medications to those approved for the study
* No heart conditions assessed by medical history and passing the PAR-Q
* Complete and pass medical exam

Exclusion Criteria:

* Positive response to any PAR-Q questions
* Physical problems/injuries associated with walking or cycling
* VO2Max below 45 ml/kg/min for men and 40 ml/kg/min for women
* Allergy to sulfa drugs
* Existing heart and or lung conditions
* Pregnant or breastfeeding
* History of heat illness or heat injury
* History of kidney stones or chronic renal problems
* History of orthostatic hypotension, diabetes or gout
* Taking certain medications: NSAIDS [anti-inflammatory/pain medications], digitalis [a type of heart medication], lithium and anti-depressants [medications used in psychiatry], anti-hypertensives [medications to lower the blood pressure], anti-fungals [medications used to treat infectious type of mold], supplements or anti-cholinergic drugs)
* Taking any supplements, particularly creatine in 24 hours before the start of the study, or during the study
* Alcohol consumption 24 hours before the start of the study, or during the study
* Incapable to give informed consent
* Anemia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Aerobically fit individuals
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Wagner, M.D., Principal Investigator — University of California, San Diego; Sarka Southern, Ph.D., Principal Investigator — Gaia Medical Institute
Locations (1):
- Clinical and Translational Research Institute, San Diego, California, United States